CLINICAL TRIAL: NCT02388035
Title: Cefotaxime Resistance in Treatment of Spontaneous Bacterial Peritonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Ahmed Ali Elbaz (Other Government)
Responsible Party: Sponsor-Investigator, Dr Ahmed Ali Elbaz, Dr, Nasser Institute For Research and Treatment
Organization: Nasser Institute For Research and Treatment (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHAEREDS-2015
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Spontaneous Bacterial Peritonitis
Keywords: profiles changes; microorganisms; cefotaxime; SBP; Egyptian; effective antibiotics
MeSH Terms: interventions — Cefotaxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SBP-group 1 (Experimental): Spontanous bacterial peritonitis
  Interventions: Drug: Cefotaxime
- CNNA-group 2 (Experimental): Culture negative neutrocytic ascites
  Interventions: Drug: Cefotaxime
- MNBA-group 3 (Experimental): monomicrobial non-neutrocytic ascites
  Interventions: Drug: Cefotaxime
- group 4 (No Intervention): no evidence of ascitic fluid infection

INTERVENTIONS:
Drug: Cefotaxime
  Arms: CNNA-group 2; MNBA-group 3; SBP-group 1

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is a serious complication in cirrhotic patients, and the changes in the microbiological characteristics reported in the last years are impacting the choice of antibiotic used in the treatment. Cefotaxime has been the most extensively studied antibiotic for this infection. It is considered to be one of the first choice antibiotics because of low toxicity and excellent efficacy. Treatment of SBP by intravenous cefotaxime should be administered for a minimum 5 days. Antibiotic-resistant microorganisms have been increasingly reported especially to cefotaxime and its effect on the clinical outcome in treating SBP.

ELIGIBILITY:
Inclusion Criteria:

* patients with liver cirrhosis and ascites and clinical findings suspicious of ascitic fluid infection

Exclusion Criteria:

* Patients were excluded if they received antibiotics ten days prior to the hospital admission or there is evidence of secondary bacterial peritonitis, tuberculous peritonitis, malignant ascites or ascites due to other causes e.g. cardiac or renal diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Organisms detected with their antibiotics sensitivity | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nasser institute, Cairo, Shubra, Egypt